CLINICAL TRIAL: NCT05777213
Title: Effectiveness of Giving Injection of Human Umbilical Cord Secretome in the Case of Trophic Ulcers (Pre-post Intervention)
Brief Title: Potential Injection of Human Umbilical Cord Secretome in the Case of Trophic Ulcers (Pre-post Intervention)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yohanes Firmansyah, dr, MH, MM (Other)
Collaborators: Tarumanagara University (Other)
Responsible Party: Sponsor-Investigator, Yohanes Firmansyah, dr, MH, MM, Researcher, Tarumanagara University
Organization: Tarumanagara University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPZ20192072
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: CM-MSC ; Stem Cell ; Trophic Ulcer ; Leprosy ; Morbun Hansen; Secretom
MeSH Terms: conditions — Leprosy | interventions — Secretome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Conditioned Medium Wharton's Jelly-derived mesenchymal stem cells (CM-WJMSCs) (Experimental): Conditioned Medium Wharton's Jelly-derived mesenchymal stem cells (CM-WJMSCs) made as much as 0.1cc / 1cm intracutaneously with a flexpen device in the wound area every 2 weeks.
  Interventions: Biological: Secretome

INTERVENTIONS:
Biological: Secretome — The interventions given in this study were Conditioned Medium Wharton's Jelly-derived mesenchymal stem cells (CM-WJMSCs) as much as 0.1cc / 1cm intracutaneously with a flexpen device in the wound area every 2 weeks. The variables in this study were divided into two, namely the independent variable was the use of Conditioned Medium Wharton's Jelly-derived mesenchymal stem cells (CM-WJMSCs) were administered intracutaneously, and the dependent variables were wound healing and side effects caused by the interventions given. Wound healing or repair in this study was assessed from several variables, namely the presence of granulation tissue growth, reduced edema, reduced erythema and improvement in wound size both in terms of length, width, and area measured by using a standard ruler and digital photo.

SUMMARY:
Background: Trophic ulcer is one of the complications that arise due to leprosy infection of the skin and includes diseases that trigger permanent disability and reduce the quality of life of the person. The facts in the field that more than 50% of chronic ulcers, especially trophic ulcers due to leprosy fail to heal with usual treatment. Therefore it is important to do a new method in healing trophic ulcers. Stem cell therapy or one of them is conditioned medium mesenchymal stem cell is a promising therapy because of its biological and physiological processes resembling the mechanism of wound healing Method: This research is a clinical trial research "Open Trial". Phase 1 to see the side effects caused by the intervention. Minimum sample size of 20 respondents with trophic ulcers due to leprosy that is difficult to resolve with usual treatment. The main outcome is wound healing in terms of the length and extent of the wound. The secondary outcome is treatment toxicity 4 weeks after administration. Follow-up visits will be scheduled at 2, 4, and 12 weeks post-treatment. If the results confirm safety, feasibility and potential efficacy, large multicenter randomized controlled trials with longer follow-up will begin with a focus on the effectiveness of therapy

ELIGIBILITY:
Inclusion Criteria:

* Chronic ulcers in Morbus Hansen's patients aged 18-80 years
* Not recovering with routine therapy for at least 1 months
* Trophic ulcers degrees 2 and 3
* Willing to take part in the study
* As well as with the respondent's good health to follow this study.

Exclusion Criteria:

* Patients who took anticoagulants,
* Patients had hypertension
* Patients had any staging kidney failure
* Patients had a history of blood disorders and pregnancy.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Changes in Wound Size - Length | 4 weeks
  Digital measurements of Length carried out using a rule from time to time (1 time per week for 4 weeks) with units in cm
Changes in Wound Size - Width | 4 weeks
  Digital measurements of Width carried out using a rule from time to time (1 time per week for 4 weeks) with units in cm
Changes in Wound Size - Area | 4 weeks
  Digital measurements carried out by multiplying the length and width of the wound over time (1 time per week for 4 weeks) in units of cm squares

OTHER OUTCOMES:
Adverse event of Allergic | 4 weeks
  Assessment of side effects in the form of allergies for 4 weeks the intervention is expressed in the form of incidence with consideration of diagnosis by a doctor and sought to know about the causal from these side effects
Adverse event of Erythema | 4 weeks
  Assessment of side effects in the form of erythema for 4 weeks the intervention is expressed in the form of incidence with consideration of diagnosis by a doctor and searched for causal from these side effects
Adverse event of Angioedema and Urticaria | 4 weeks
  Assessment of side effects in the form of Angioedema and Urticaria for 4 weeks the intervention is expressed in the form of incidence with consideration of diagnosis by a doctor and searched for causal from these side effects
Adverse event of Tumor | 4 weeks
  Assessment of side effects in the form of Tumor for 4 weeks the intervention is expressed in the form of incidence with consideration of diagnosis by a doctor and searched for causal from these side effects

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Sukma Clinic, Tangerang, Banten
  - RS Alverno Singkawang, Singkawang, West Borneo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Santos VS, Santos LC, Lobo LV, Lemos LM, Gurgel RQ, Cuevas LE. Leprosy and disability in children younger than 15 years in an endemic area of northeast Brazil. Pediatr Infect Dis J. 2015 Mar;34(3):e44-7. doi: 10.1097/INF.0000000000000592. PMID 25389921
- [Result] Santos VS, de Matos AM, de Oliveira LS, de Lemos LM, Gurgel RQ, Reis FP, Santos VT, Feitosa VL. Clinical variables associated with disability in leprosy cases in northeast Brazil. J Infect Dev Ctries. 2015 Mar 15;9(3):232-8. doi: 10.3855/jidc.5341. PMID 25771459
- [Result] de Paula HL, de Souza CDF, Silva SR, Martins-Filho PRS, Barreto JG, Gurgel RQ, Cuevas LE, Santos VS. Risk Factors for Physical Disability in Patients With Leprosy: A Systematic Review and Meta-analysis. JAMA Dermatol. 2019 Oct 1;155(10):1120-1128. doi: 10.1001/jamadermatol.2019.1768. PMID 31389998
- [Result] van Brakel WH, Sihombing B, Djarir H, Beise K, Kusumawardhani L, Yulihane R, Kurniasari I, Kasim M, Kesumaningsih KI, Wilder-Smith A. Disability in people affected by leprosy: the role of impairment, activity, social participation, stigma and discrimination. Glob Health Action. 2012;5. doi: 10.3402/gha.v5i0.18394. Epub 2012 Jul 20. PMID 22826694
- [Result] Gahalaut P, Pinto J, Pai GS, Kamath J, Joshua TV. A novel treatment for plantar ulcers in leprosy: local superficial flaps. Lepr Rev. 2005 Sep;76(3):220-31. PMID 16248209
- [Result] Pawitan JA. Prospect of stem cell conditioned medium in regenerative medicine. Biomed Res Int. 2014;2014:965849. doi: 10.1155/2014/965849. Epub 2014 Aug 28. PMID 25530971
- [Result] Li CY, Wu XY, Tong JB, Yang XX, Zhao JL, Zheng QF, Zhao GB, Ma ZJ. Comparative analysis of human mesenchymal stem cells from bone marrow and adipose tissue under xeno-free conditions for cell therapy. Stem Cell Res Ther. 2015 Apr 13;6(1):55. doi: 10.1186/s13287-015-0066-5. PMID 25884704
- [Result] Sarasua JG, Lopez SP, Viejo MA, Basterrechea MP, Rodriguez AF, Gutierrez AF, Gala JG, Menendez YM, Augusto DE, Arias AP, Hernandez JO. Treatment of pressure ulcers with autologous bone marrow nuclear cells in patients with spinal cord injury. J Spinal Cord Med. 2011;34(3):301-7. doi: 10.1179/2045772311Y.0000000010. PMID 21756569
- [Result] Vizoso FJ, Eiro N, Cid S, Schneider J, Perez-Fernandez R. Mesenchymal Stem Cell Secretome: Toward Cell-Free Therapeutic Strategies in Regenerative Medicine. Int J Mol Sci. 2017 Aug 25;18(9):1852. doi: 10.3390/ijms18091852. PMID 28841158
- [Result] Natallya FR, Herwanto N, Prakoeswa C, Indramaya DM, Rantam FA. Effective Healing of Leprosy Chronic Plantar Ulcers by Application of Human Amniotic Membrane Stem Cell Secretome Gel. Indian J Dermatol. 2019 May-Jun;64(3):250. doi: 10.4103/ijd.IJD_6_17. PMID 31148869
- [Result] Liew A, O'Brien T. Therapeutic potential for mesenchymal stem cell transplantation in critical limb ischemia. Stem Cell Res Ther. 2012 Jul 30;3(4):28. doi: 10.1186/scrt119. PMID 22846185